CLINICAL TRIAL: NCT05601804
Title: TARGETing Healthy Weight Loss in the Context of Food Insecurity Pilot and Feasibility Trial I
Brief Title: TARGETing Healthy Weight Loss in the Context of Food Insecurity
Acronym: TARGET P&F I
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Candice A. Myers, Ph.D., Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2022-039
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Food Insecurity; Food Security; Body Weight
Keywords: Food Insecurity; Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Food Insecure Women with Obesity: 4 focus groups with 6-8 participants each
- Food Secure Women with Obesity: 3 focus groups with 6-8 participants each

SUMMARY:
This pilot and feasibility study will collect information from food insecure, as well as food secure, women with obesity to detail their desires and needs for healthy weight reduction. Up to 60 women with obesity will be enrolled. Pennington Biomedical Research Center will coordinate this qualitative study and use focus groups discussion to collect formative data.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Female
* 18 to 65 years of age
* BMI ≥ 30 kg/m2
* Ability to read and write using English
* Willing to participate in focus group discussions
* Willing to be audio/video recorded

Exclusion Criteria:

* Male
* Currently pregnant
* BMI <30 kg/m2

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 to 65 years with a BMI of 30.0 kg/m2 or greater.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Desires and needs for weight loss | Through study completion, up to 1 year
  Via focus group discussions, we will elicit in-depth information from women with food insecurity and obesity to detail their desires and needs for weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Candice A. Myers, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States